CLINICAL TRIAL: NCT02659631
Title: A PHASE 1 DOSE ESCALATION STUDY EVALUATING THE SAFETY AND TOLERABILITY OF PF-06671008 IN PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: PF-06671008 Dose Escalation Study in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7831001
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Neoplasms
Keywords: P-cadherin; PF-06671008; solid tumors; lung cancer; breast cancer; colorectal cancer; NSCLC; TNBC; CRC; neoplasms; Triple negative breast cancer; Non-small cell lung cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — PF-06671008

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-06671008 (Experimental)
  Interventions: Drug: PF-06671008

INTERVENTIONS:
Drug: PF-06671008 — Dose Escalation Phase - Part 1
Drug: PF-06671008 — Dose Expansion Phase - Part 2

SUMMARY:
The study will evaluate the safety, pharmacokinetics and pharmacodynamics of increasing doses of PF-06671008 in patients with advanced solid tumors with the potential to have P-cadherin expression. The study will then expand to look at the selected dose in patients with P-cadherin expressing TNBC, CRC or NSCLC.

ELIGIBILITY:
Key Inclusion Criteria

* Diagnosis of tumor type with the potential to have P-cadherin expression that is resistant to standard therapy or for which no standard therapy is available
* Performance status of 0 or 1
* Adequate bone marrow, kidney and liver function

Key Exclusion Criteria

* Known CNS disease including, but not limited to, metastases
* Current or history of seizure disorder
* History of or active autoimmune disorders
* Active bacterial, fungal or viral infection
* Major surgery, anti-cancer therapy, or radiation therapy within 4 weeks of study treatment
* Requirement for systemic immune suppressive medication
* Grade 2 or greater peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Memorial Sloan Kettering Cancer Center - Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center- Clinical Trials Office, New York, New York
  - Memorial Sloan Kettering Cancer Center Rockefeller Outpatient Pavillion, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The University of Texas - M.D. Anderson Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Harding JJ, Garrido-Laguna I, Chen X, Basu C, Dowlati A, Forgie A, Hooper AT, Kamperschroer C, Max SI, Moreau A, Shannon M, Wong GY, Hong DS. A Phase 1 Dose-Escalation Study of PF-06671008, a Bispecific T-Cell-Engaging Therapy Targeting P-Cadherin in Patients With Advanced Solid Tumors. Front Immunol. 2022 Apr 14;13:845417. doi: 10.3389/fimmu.2022.845417. eCollection 2022. PMID 35493516
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7831001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-eight (28) participants were enrolled and 27 participants received study drug. One participant discontinued before receiving treatment.
Groups:
- PF-06671008 1.5 ng/kg IV: PF-06671008 was administered as a weekly intravenous (IV) infusion in 21-day cycles at 1.5 nanogram/kilogram (ng/kg). PF-06671008 was administered for up to 4 cycles in this cohort.
- PF-06671008 7.5 ng/kg IV: PF-06671008 was administered as a weekly IV infusion in 21-day cycles at 7.5 ng/kg. PF-06671008 was administered for up to 3 cycles in this cohort.
- PF-06671008 20 ng/kg IV: PF-06671008 was administered as a weekly IV infusion in 21-day cycles at 20 ng/kg. PF-06671008 was administered for up to 4 cycles in this cohort.
- PF-06671008 50 ng/kg IV: PF-06671008 was administered as a weekly IV infusion in 21-day cycles at 50 ng/kg. PF-06671008 was administered for up to 2 cycles in this cohort.
- PF-06671008 100 ng/kg IV: PF-06671008 was administered as a weekly IV infusion in 21-day cycles at 100 ng/kg. PF-06671008 was administered for up to 4 cycles in this cohort.
- PF-06671008 200 ng/kg IV: PF-06671008 was administered as a weekly IV infusion in 21-day cycles at 200 ng/kg. PF-06671008 was administered for up to 16 cycles in this cohort.
- PF-06671008 300 ng/kg IV: PF-06671008 was administered as a weekly IV infusion in 21-day cycles at 300 ng/kg. PF-06671008 was administered for up to 4 cycles in this cohort.
- PF-06671008 400 ng/kg IV: PF-06671008 was administered as a weekly IV infusion in 21-day cycles at 400 ng/kg. PF-06671008 was administered for up to 2 cycles in this cohort.
- PF-06671008 200 ng/kg SC: PF-06671008 was administered as a weekly subcutaneous (SC) injection in 21-day cycles at 200 ng/kg. PF-06671008 was administered for up to 5 cycles in this cohort.
- PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV: PF-06671008 was administered as a weekly IV infusion in 21-day cycles at a priming dose of 200 ng/kg on Cycle 1 Day 1 (C1D1) and 300 ng/kg for all subsequent dosing. PF-06671008 was administered for up to 4 cycles in this cohort.
Period: Overall Study
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Started (This study was terminated early and Part 2 was not initiated. The form only includes arms in Part 1.) | 1 | 2 | 3 | 2 | 5 | 5 | 4 | 3 | 2 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1
Not Completed | 1 | 2 | 3 | 2 | 5 | 3 | 1 | 3 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal prior to treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant refused further follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death (follow-up phase) | 1 | 2 | 1 | 1 | 3 | 2 | 0 | 3 | 1 | 0
Not completed — Death (treatment phase) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants treated (27)
Groups:
- PF-06671008 1.5 ng/kg IV: PF-06671008 was administered as a weekly intravenous (IV) infusion in 21-day cycles at 1.5 ng/kg. PF-06671008 was administered for up to 4 cycles in this cohort.
- Total: Total of all reporting groups
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV | Total
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1 | 27
Age, Customized [Number; unit: Participants]
  < 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 44 years | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 6
  45 - 64 years | 1 | 2 | 2 | 0 | 0 | 3 | 1 | 2 | 0 | 1 | 12
  ≥ 65 years | 0 | 0 | 0 | 1 | 4 | 1 | 2 | 1 | 0 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 1 | 4 | 0 | 1 | 1 | 0 | 12
  Male | 1 | 1 | 1 | 0 | 3 | 1 | 4 | 2 | 1 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 1 | 2 | 2 | 2 | 4 | 4 | 4 | 3 | 2 | 1 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 1 | 3 | 2 | 3 | 3 | 3 | 2 | 2 | 1 | 21
  Black | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 4
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) - Part 1
Description: DLT was defined as any of the following adverse events occurring in the first cycle of treatment (21 days after the first dose): a) Hematologic: Febrile neutropenia defined as an absolute neutrophil count (ANC) <1.0 x 10^9/L with a single temperature of >38.3°C, or 101°F, or a sustained temperature of >=38°C, or 100.4°F, for more than one hour; b) Non-hematologic: Delay by more than 2 weeks in receiving the next scheduled dose due to persisting treatment related toxicities; c) Any grade 3 or 4 clinically-relevant hematologic or non-hematologic toxicity.
Time Frame: Baseline through Day 21 (Cycle 1)
Population: All enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Objective Response (OR) - Part 2
Description: Number of participants with OR based on assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) v1.1.
  CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions.
  PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months
Population: This study was terminated early and Part 2 was not initiated. Data for this outcome measure was not collected.
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Serum Concentration (Cmax) of PF-06671008
Description: Maximum serum concentration (Cmax) of PF-06671008 was observed directly from data.
  Geometric mean was not calculated if fewer than 3 participants had reportable parameter values.
Time Frame: C1D1 0, 1, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose, C2D1 0, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose
Population: All enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest and who had no major protocol deviations influencing the PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
nanogram/milliliter (ng/mL)
  Cycle 1 Day 1 | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 0.1926 (20) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 1.108 (32) | 2.008 (33) | 2.387 (36) | 4.049 (14) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values.
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 1 | 3 | 4 | 2 | 0 | 2 | 1
  Cycle 2 Day 1 | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 0.2470 (36) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 0.8471 (51) | 2.014 (7) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. |  | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values.

4. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-06671008
Description: Time for Maximum serum concentration (Tmax) of PF-06671008 was observed directly from data as time of first occurrence.
Time Frame: C1D1 0, 1, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose, C2D1 0, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
hours
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
  Cycle 1 Day 1 |  | 2.02 [2.02 to 2.02] | 4.05 [2.00 to 4.08] | 2.29 [1.92 to 2.65] | 2.07 [2.00 to 4.10] | 2.33 [2.00 to 3.98] | 2.17 [2.05 to 3.63] | 2.05 [2.05 to 3.00] | 50.5 [8.12 to 92.9] | 1.92 [1.92 to 1.92]
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 1 | 3 | 4 | 2 | 0 | 2 | 1
  Cycle 2 Day 1 |  | 2.12 [2.12 to 2.12] | 3.98 [2.00 to 4.22] | 3.90 [3.90 to 3.90] | 4.00 [2.17 to 4.28] | 2.09 [1.92 to 2.17] | 2.14 [2.10 to 2.17] |  | 24.6 [23.4 to 25.7] | 1.98 [1.98 to 1.98]

5. Secondary Outcome: Terminal Elimination Half-life (t1/2) of PF-06671008
Description: Terminal elimination half-life (t1/2) of PF-06671008 was calculated as ln(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
  Arithmetic mean was not calculated if fewer than 3 participants had reportable parameter values.
Time Frame: C1D1 0, 1, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose, C2D1 0, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
hours
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 3 | 2 | 2 | 0 | 1
  Cycle 1 Day 1 |  |  |  | NA (NA) — Summary statistics are not presented as arithmetic means were not calculated if fewer than 3 participants had reportable values. | 31.77 (7.6055) | 35.30 (5.4065) | NA (NA) — Summary statistics are not presented as arithmetic means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as arithmetic means were not calculated if fewer than 3 participants had reportable values. |  | NA (NA) — Summary statistics are not presented as arithmetic means were not calculated if fewer than 3 participants had reportable values.
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
  Cycle 2 Day 1 |  |  |  |  | NA (NA) — Summary statistics are not presented as arithmetic means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as arithmetic means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as arithmetic means were not calculated if fewer than 3 participants had reportable values. |  |  |

6. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06671008
Description: Tau refers to the dosing interval, which was 1 week. Area under the concentration-time profile from time 0 to time tau (AUCtau) was determined using linear/log trapezoidal method.
  Geometric mean was not calculated if fewer than 3 participants had reportable parameter values.
Time Frame: C1D1 0, 1, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose, C2D1 0, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram.hour/milliliter (ng.hr/mL)
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
nanogram.hour/milliliter (ng.hr/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 2 | 2 | 2 | 1
  Cycle 1 Day 1 | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 5.252 (25) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 42.75 (35) | 87.31 (29) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values.
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 1 | 1 | 3 | 1 | 0 | 2 | 1
  Cycle 2 Day 1 | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 10.31 (43) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 79.17 (36) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. |  | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values.

7. Secondary Outcome: Area Under the Curve From Time 0 Extrapolated to Infinity Time (AUCinf) of PF-06671008
Description: AUCinf was calculated as AUClast +(Clast*/kel), where AUClast is area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* is the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis, kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
  Geometric mean was not calculated if fewer than 3 participants had reportable parameter values.
Time Frame: C1D1 0, 1, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose, C2D1 0, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
ng.hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 3 | 2 | 2 | 0 | 1
  Cycle 1 Day 1 |  |  |  | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 47.09 (41) | 90.35 (19) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. |  | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values.
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Systemic Clearance (CL) of PF-06671008
Description: Systemic Clearance (CL) was calculated as dose/AUCinf, where AUCinf was area under the serum concentration-time profile from time 0 extrapolated to infinite time. This outcome measure only applies to IV arms.
  Geometric mean was not calculated if fewer than 3 participants had reportable parameter values.
Time Frame: C1D1 0, 1, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose, C2D1 0, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/hour/kilogram (mL/hr/kg)
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 1
milliliter/hour/kilogram (mL/hr/kg)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 3 | 2 | 2 | 1
  Cycle 1 Day 1 |  |  |  | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 2.191 (47) | 2.236 (20) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values.
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 1 | 1 | 3 | 1 | 0 | 1
  Cycle 2 Day 1 |  | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 1.954 (40) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. | 1.827 (77) | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values. |  | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values.

9. Secondary Outcome: Apparent Clearance (CL/F) of PF-06671008
Description: Apparent Clearance (CL/F) was calculated as dose/AUCinf, where AUCinf was area under the serum concentration-time profile from time 0 extrapolated to infinite time. This outcome measure only applies to SC arm.
  Geometric mean was not calculated if fewer than 3 participants had reportable parameter values.
Time Frame: C1D1 0, 1, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose, C2D1 0, 2, 4, 8, 24, 48, 72 and 96 hrs post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | PF-06671008 200 ng/kg SC
Number analyzed (Participants) | 2
mL/hr/kg
  Cycle 1 Day 1: number analyzed (Participants) | 0
  Cycle 2 Day 1 | NA (NA) — Summary statistics are not presented as geometric means were not calculated if fewer than 3 participants had reportable values.

10. Secondary Outcome: Number of Participants With OR - Part 1
Description: Number of participants with OR based on assessment of CR or PR according to RECIST v1.1.
  CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions.
  PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline and every 6 weeks for the first 6 months, then every 12 weeks until disease progression, unacceptable toxicity, or up to 24 months
Population: All randomized participants who received at least 1 dose of study intervention, had measurable disease baseline assessment and at least 1 post baseline assessment or disease progression or death before the first tumor assessment. No participants met the criteria of OR.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) - Part 2
Description: The period from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline and every 6 weeks for the first 6 months, then every 12 weeks until disease progression or unacceptable toxicity, or up to 24 months
Population: This study was terminated early and Part 2 was not initiated. Data for this outcome measure were not collected.
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Overall Survival (OS) - Part 2
Description: The period from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 7. Death was determined from AE data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: as for outcome 11
Population: This study was terminated early and Part 2 was not initiated. Data for this outcome measure were not collected.
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Anti Drug Antibodies (ADA) and Neutralizing Antibodies (NAb) Against PF-06671008
Description: ADA against PF-06671008 in human serum samples was determined following a tiered approach using screening, confirmation, and titer/quantification by semi-quantitative enzyme linked immunosorbent assay (ELISA). Endpoint titer >=1.18 was considered positive.
Time Frame: C1D1 0 hrs, D15 0 hrs, and C2D1 0 hrs, and D1 0 hrs post additional dosings, up to 24 months
Population: All enrolled participants who received at least one dose of study intervention and had at least one post dose ADA sample analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 5 | 4 | 3 | 2 | 1
Participants
  ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  NAb | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study. | NA — NAb samples were not analyzed for this study.

ADVERSE EVENTS:
Time Frame: For all Adverse Events: Start of treatment to and including 28 days after the last dose. For All-Cause Mortality: Start of treatment to and including 28 days after the last dose + follow-up period (up to 2 years)
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-06671008 1.5 ng/kg IV | PF-06671008 7.5 ng/kg IV | PF-06671008 20 ng/kg IV | PF-06671008 50 ng/kg IV | PF-06671008 100 ng/kg IV | PF-06671008 200 ng/kg IV | PF-06671008 300 ng/kg IV | PF-06671008 400 ng/kg IV | PF-06671008 200 ng/kg SC | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV
All-Cause Mortality (participants affected / at risk) | 1/1 | 2/2 | 1/3 | 1/2 | 4/4 | 2/5 | 1/4 | 3/3 | 1/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 1/3 | 2/2 | 4/4 | 4/5 | 3/4 | 2/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 3/3 | 2/2 | 4/4 | 5/5 | 4/4 | 3/3 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06671008 1.5 ng/kg IV (N=1) | PF-06671008 7.5 ng/kg IV (N=2) | PF-06671008 20 ng/kg IV (N=3) | PF-06671008 50 ng/kg IV (N=2) | PF-06671008 100 ng/kg IV (N=4) | PF-06671008 200 ng/kg IV (N=5) | PF-06671008 300 ng/kg IV (N=4) | PF-06671008 400 ng/kg IV (N=3) | PF-06671008 200 ng/kg SC (N=2) | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 2 | 4 | 4 | 3 | 2 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06671008 1.5 ng/kg IV (N=1) | PF-06671008 7.5 ng/kg IV (N=2) | PF-06671008 20 ng/kg IV (N=3) | PF-06671008 50 ng/kg IV (N=2) | PF-06671008 100 ng/kg IV (N=4) | PF-06671008 200 ng/kg IV (N=5) | PF-06671008 300 ng/kg IV (N=4) | PF-06671008 400 ng/kg IV (N=3) | PF-06671008 200 ng/kg SC (N=2) | PF-06671008 200 ng/kg Prime and 300 ng/kg Maintenance IV (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 1 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 3 | 2 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 1 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT02659631/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT02659631/SAP_001.pdf